CLINICAL TRIAL: NCT00660283
Title: A Phase II Study of Gliadel, Concomitant Temozolomide and Radiation, Followed By Dose Dense Therapy With Temozolomide For Newly Diagnosed Malignant High Grade Glioma
Acronym: KARE003
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Kentuckiana Cancer Institute (Other)
Collaborators: Eisai Inc. (Industry)
Responsible Party: Renato V. LaRocca, MD, Kentuckiana Cancer Institute
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: KARE003; KARE 003
Record Dates: First submitted 2008-04-14; First posted 2008-04-17 (Estimated); Last update posted 2010-01-20 (Estimated); Status verified 2010-01

CONDITIONS: Glioma
Keywords: GBM; Newly; diagnosed; malignant; high grade
MeSH Terms: conditions — Glioma; Disease | interventions — Temozolomide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: Temozolomide — (Stage I Treatment) Postoperative concomitant limited-field radiation therapy with daily temozolomide (75 mg/m2) must begin between 14 and 28 days from surgery.
  7. (Stage II Treatment) temozolomide 150 mg/m2 to be given days 1-7 and 15-21 of a 28 day cycle to begin within 45 days of stop date of concomitant limited field radiation/daily temozolomide (Stage I treatment) up to a maximum of 12 cycles.

SUMMARY:
To determine the safety and efficacy of surgical resection with Gliadel® 3.85% wafer implantation, followed by concomitant limited field radiation therapy and temozolomide, followed by dose dense temozolomide in subjects undergoing initial surgery for newly-diagnosed high grade glioma.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects, men and women, must be between ages 18 and 75 years.
2. Subjects must have radiographic evidence on cranial magnetic resonance imaging (MRI) of a single, contrast-enhancing unilateral supratentorial cerebral tumor (see Section 8.4).

3 Surgery is recommended within 4 weeks of the baseline MRI scan.

4. Subjects must have a Karnofsky Performance Score of 60 or higher.

5. Subjects must have signed an Institutional Review Board (IRB)-approved informed consent prior to any non-standard of care study procedure or no later than the start of dose dense temozolomide.

6. Subjects must have a pathological diagnosis of a high grade (IV) malignant glioma.

7. Subjects, both men and women, must be willing to avoid pregnancy for up to 2 years after wafer implantation surgery and be counseled regarding the unknown, and potentially harmful, risks to the embryo or fetus from participation in this study.

Exclusion Criteria:

1. Subjects who have had prior cytoreductive surgery for high-grade glioma. Subjects who have had a diagnostic stereotactic biopsy are eligible.
2. Subjects with more than one focus of tumor or tumor crossing the midline as assessed by coronal cranial MRI scan.
3. Concomitant significant life-threatening disease from which the subject could reasonably be expected to die within the first 12 months of the study.
4. Known hypersensitivity reactions to temozolomide, nitrosoureas or any other components of the Gliadel® wafer.
5. Prior CNS radiotherapy.
6. Subjects who have received any prior chemotherapy for this malignant glioma prior to the baseline evaluation or subjects who are currently being treated with chemotherapeutic agents.
7. Subjects with fewer than 100,000 platelets per mm3 or fewer than 3.500 leukocytes per mm3.
8. Liver function tests greater than or equal to 2.5 times the upper limit of normal (transaminases (SGOT, SGPT), total bilirubin, alkaline phosphatase).
9. Serum creatinine equal to or greater than 1.5 times the upper limit of normal, blood urea nitrogen (BUN) equal to or greater than 2.5 times the upper limit of normal.
10. Pregnancy, or lactating females or females of childbearing potential not using adequate contraception.
11. Participation in any other investigational protocol in the prior twelve months for any type of malignancy.
12. Psychological, familial, sociological or geographical conditions which do not permit adequate medical follow-up and compliance with the study protocol.
13. Inadequately controlled hypertension (blood pressure systolic > 150 mmHg or diastolic > 100 mmHg).
14. Unstable angina or history of myocardial infarction within six months prior to enrollment.
15. Evidence of bleeding, diathesis, or coagulopathy. Chronic full-dose anticoagulation with warfarin is not permitted though subjects may be on low molecular weight heparin or fondaparinux.
16. Serious non-healing wound, ulcer, or bone fracture.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2009-01; Primary Completion 2010-12 (Estimated); Study Completion 2010-12 (Estimated)

PRIMARY OUTCOMES:
Safety and efficacy of concomitant limited field radiation therapy and temozolomide, followed by dose dense temozolomide in subjects undergoing initial surgery for newly-diagnosed high grade glioma. | 1st five subjects at 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Renato V LaRocca, MD, Principal Investigator — Kentuckiana Cancer Instititue
Locations (1):
- Kentuckiana Cancer Institute, Louisville, Kentucky, United States